CLINICAL TRIAL: NCT05074368
Title: Comparative Analysis of Neutralizing Antibody Response Among Heterologous ChAdOx1-nCov-19/mRNA-1273 Vaccination and Homologous ChAdOx1-nCov-19 or Homologous mRNA-1273 Vaccination
Brief Title: Efficacy and Safety of Heterologous and Homologous COVID-19 Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Taoyuan General Hospital, Ministry of Health and Welfare,Taoyuan,Taiwan (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202106039MINA
Record Dates: First submitted 2021-08-24; First posted 2021-10-12 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2021-10

CONDITIONS: Healthy Adult Volunteers
Keywords: adenovirus-vector ChAdOx1 vaccination; messenger RNA (mRNA-1273 )vaccination; Coronavirus disease 2019 (COVID-19); humoral immunity; SARS-CoV-2; adverse events
MeSH Terms: conditions — COVID-19 | interventions — ChAdOx1 nCoV-19; Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Heterologous ChAdOx1-nCov-19 vaccination - 8 weeks apart (Active Comparator): Astra-Zeneca vaccine 0.5 mL/dose
  Interventions: Biological: ChAdOx1-nCov-19 (Astra-Zeneca)
- mRNA-1273 Vaccination and Heterologous ChAdOx1-nCov-19 vaccination- 8 weeks apart (Active Comparator): Moderna COVID-19 Vaccine 0.5 mL/dose and Astra-Zeneca vaccine 0.5 mL/dose
  Interventions: Biological: ChAdOx1-nCov-19 (Astra-Zeneca); Biological: SARS-CoV-2 messenger RNA-1273 (Moderna) vaccine
- Heterologous ChAdOx1-nCov-19 vaccination and the mRNA-1273 Vaccination- 4 weeks apart (Active Comparator): Moderna COVID-19 Vaccine 0.5 mL/dose and Astra-Zeneca vaccine 0.5 mL/dose
  Interventions: Biological: ChAdOx1-nCov-19 (Astra-Zeneca); Biological: SARS-CoV-2 messenger RNA-1273 (Moderna) vaccine
- The mRNA-1273 Vaccination- 4 weeks apart (Active Comparator): Moderna COVID-19 Vaccine 0.5 mL/dose
  Interventions: Biological: SARS-CoV-2 messenger RNA-1273 (Moderna) vaccine
- Heterologous ChAdOx1-nCov-19 vaccination and the mRNA-1273 Vaccination-12 weeks apart (Active Comparator): Moderna COVID-19 Vaccine 0.5 mL/dose and Astra-Zeneca vaccine 0.5 mL/dose
  Interventions: Biological: ChAdOx1-nCov-19 (Astra-Zeneca); Biological: SARS-CoV-2 messenger RNA-1273 (Moderna) vaccine

INTERVENTIONS:
Biological: ChAdOx1-nCov-19 (Astra-Zeneca) — vaccine inoculation and mixed inoculation
  Arms: Heterologous ChAdOx1-nCov-19 vaccination - 8 weeks apart; Heterologous ChAdOx1-nCov-19 vaccination and the mRNA-1273 Vaccination- 4 weeks apart; Heterologous ChAdOx1-nCov-19 vaccination and the mRNA-1273 Vaccination-12 weeks apart; mRNA-1273 Vaccination and Heterologous ChAdOx1-nCov-19 vaccination- 8 weeks apart
Biological: SARS-CoV-2 messenger RNA-1273 (Moderna) vaccine — vaccine inoculation and mixed inoculation
  Arms: Heterologous ChAdOx1-nCov-19 vaccination and the mRNA-1273 Vaccination- 4 weeks apart; Heterologous ChAdOx1-nCov-19 vaccination and the mRNA-1273 Vaccination-12 weeks apart; The mRNA-1273 Vaccination- 4 weeks apart; mRNA-1273 Vaccination and Heterologous ChAdOx1-nCov-19 vaccination- 8 weeks apart

SUMMARY:
The investigators conduct a prospective analysis to compare homologous and heterologous adenovirus vector ChAdOx1-nCov-19 (Astra-Zeneca) or SARS-CoV-2 messenger RNA-1273 (Moderna) vaccine inoculation. Healthy volunteers will be enrolled and divided into five groups. The first group is the subjects who received ChAdOx1- nCov-19 vaccine with 8 weeks apart; the second group is the SARS-CoV-2 messenger RNA-1273 vaccine after the first dose of ChAdOx1-nCov-19 vaccination with 8 weeks apart; the third group is the first dose of ChAdOx1-nCov-19 vaccine and the SARS-CoV-2 messenger RNA-1273 vaccine with 4 weeks apart; the fourth group is the SARS-CoV-2 messenger RNA-1273 vaccination with 4 weeks apart; the fifth group is the first dose of ChAdOx1-nCov-19 vaccine and the SARS-CoV-2 messenger RNA-1273 vaccine with 12 weeks apart. There will be 100 volunteers in each group. Antibody test on the day before and the 14th, 28th day and 12th week after the second dose of vaccination, including 100 subjects in each group for SARS-CoV-2 ELISA antibody titer and 50 people in each group for SARS-CoV-2 neutralizing antibody titer. Adverse reactions at the first day, the 14th day, the 28th day, and the 12th week. The research team follow up each volunteer at the 6th month.

DETAILED DESCRIPTION:
The investigators would like to conduct a prospective analysis to compare the same adenovirus vector ChAdOx1-nCov-19 (Astra-Zeneca) or SARS-CoV-2 messenger RNA-1273 (Moderna) vaccine inoculation and mixed inoculation of ChAdOx1-nCov-19 and messenger RNA-1273 vaccine. Healthy volunteers (including medical personnel) will be enrolled and divided into five groups according to their wishes. The five groups are: the first group is the subjects who received ChAdOx1- nCov-19 vaccine with 8 weeks apart; the second group is the SARS-CoV-2 messenger RNA-1273 vaccine after the first dose of ChAdOx1-nCov-19 vaccination with 8 weeks apart; the third group is the first dose of ChAdOx1-nCov-19 vaccine and the SARS-CoV-2 messenger RNA-1273 vaccine with 4 weeks apart; the fourth group is the SARS-CoV-2 messenger RNA-1273 vaccination with 4 weeks apart; the fifth group is the first dose of ChAdOx1-nCov-19 vaccine and the SARS-CoV-2 messenger RNA-1273 vaccine with 12 weeks apart. There will be 100 volunteers in each group, and blood will be drawn for antibody test on the day before and the 14th, 28th day and 12th week after the second dose of vaccination, including 100 subjects in each group for SARS-CoV-2 ELISA antibody titer and 50 people in each group for SARS-CoV-2 neutralizing antibody titer. This study analyzo the titers of SARS-CoV-2 antibodies, and records adverse reactions at each visits including the first day, the 14th day, the 28th day, and the 12th week (including those within 7 days after the inoculation). Adverse reactions and whether there is development of COVID-19 within 6 months will be recorded. The research team will also follow up by phone in the 6th month to ask whether there is vaccine associated adverse events or SARS-CoV-2 infection. The results will provide information for vaccine policy in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged ≥20 to <65 years old and have received adenovirus vector vaccine ChAdOx1-nCov-19 (Astra-Zeneca) or SARS-CoV-2 messenger RNA-1273 once within three months at least four weeks apart.
2. The subject must sign the subject's inform consent, or the subject's legal representative must understand and agree, then sign inform consent according to procedure above.
3. Healthy or existing medical condition is stable, and within 3 months before being included in the trial, he or she has not been hospitalized due to illness, and his or her condition is expected to remain stable during the trial period.

Exclusion Criteria:

1. Are currently pregnant or breastfeeding or plan to become pregnant within 30 days after the second dose of the trial vaccine.
2. Currently receiving or receiving other vaccines, including Streptococcus pneumoniae vaccine.
3. Have used any blood products or intravenous immunoglobulin within 12 weeks before entering the test. Receive concurrent immunosuppressive or immunomodulatory therapy (including steroid prednisone, targeted drugs such as infliximab, adalimumab, etanercept) within 12 weeks.
4. Immunosuppressive diseases or immune insufficiency states, including hematological malignancies, parenchymal organs, bone marrow transplant history or asplenia, autoimmune diseases (systemic lupus, rheumatoid arthritis, scleroderma, polyarthritis, autoimmune thyroiditis, etc.) and human immunodeficiency virus infection.
5. Bleeding disease and assessed as a contraindication to prohibit the use of intramuscular injection or blood draw.
6. Other condition, such as physical examination or instability according to the trial investigator's judgment, or participation in this trial may adversely affect the safety of subjects, fail to comply with trial regulations, or interfere with trial evaluation indicators.
7. The subject is known to have been infected with severe acute respiratory syndrome coronavirus type 2 (SARS-CoV-2).

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Both gender allowed
Enrollment: 499 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-05-18 (Actual)

PRIMARY OUTCOMES:
Serum Samples for by using enzyme-linkes immuno sorbent assay (ELISA) at 14th,28th,12 th week and 6 months after the second dose. | 1 years
  Neutralizing antibody response among heterologous and heterologous COVID-19 vaccination and homologous

SECONDARY OUTCOMES:
Blood Sample for spike-specific CD4+ T cells | 6 months
Blood Sample for production of interferon(IFN)-γ | 6 months
  (pg/mL)
Blood Sample for tumor necrosis factor (TNF)-α | 6 months
  (pg/mL)

OTHER OUTCOMES:
Adverse events | 6 months
  Adverse events and severe adverse events at 14th,28th,12 th week and 6months after the second dose.
severe adverse events | 6 months
  Adverse events and severe adverse events at 14th,28th,12 th week and 6months after the second dose.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, X, Taiwan

REFERENCES:
- [Derived] Sheng WH, Chang SY, Lin PH, Hsieh MJ, Chang HH, Cheng CY, Yang HC, Pan CF, Ieong SM, Chao TL, Chen JP, Cheng SH, Chang SC. Immune response and safety of heterologous ChAdOx1-nCoV-19/mRNA-1273 vaccination compared with homologous ChAdOx1-nCoV-19 or homologous mRNA-1273 vaccination. J Formos Med Assoc. 2022 Apr;121(4):766-777. doi: 10.1016/j.jfma.2022.02.020. Epub 2022 Mar 16. PMID 35305895